CLINICAL TRIAL: NCT05987800
Title: Non-invasive Ventilation in Preterm Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIV study
Record Dates: First submitted 2022-11-02; First posted 2023-08-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Premature Birth; Respiratory Distress Syndrome; Ventilator Lung; Newborn
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preterm infants on non-invasive respiratory support (Other): All infants on non-invasive respiratory support will be studied. Only infants on less than 32 weeks of gestation at birth, will undergo an intervention.
  Interventions: Diagnostic Test: Titration procedure; Diagnostic Test: Electrical impedance tomography; Diagnostic Test: Lung and diaphragm ultrasound

INTERVENTIONS:
Diagnostic Test: Titration procedure — The NAVA level will be reduced to 0,5 cmH2O/microvolt (µV) for 3 minutes as a starting point. Limit peak pressure will be set to 35 cmH2O (the maxi-mum pressure that can be delivered to the patient is cut off at 30 cmH2O). Other ventilator settings will be left unchanged and are as clinically indicated.
  Starting from a NAVA level of 0,5 cmH20/µV the level will be increased by 0,5 cmH2O/µV every 3 minutes until reaching a maximum NAVA level of 2,5 cmH2O/µV.
Diagnostic Test: Electrical impedance tomography — This is a non-invasive technique consisting of the application of a non-adhesive single-use patient belt to monitor regional changes in lung aeration at the bedside.
Diagnostic Test: Lung and diaphragm ultrasound — Lung ultrasound is a non-invasive technique used to diagnose lung pathology and to monitor lung condition. This technique is part of the standard of care for preterm infants in our neonatal unit. Lung ultrasound scores are calculated at each time an ultrasound is performed.
  Ultrasound of the diaphragm consists of a short additional measurement of diaphragm thickness and thickening fraction and will be done at the same time of the lung ultrasound following a standardized procedure.

SUMMARY:
This is a prospective, observational cohort study. For the study part on noninvasive neurally adjusted ventilatory assist (NIV-NAVA) the design is interventional. For all participants prospective data collection will be conducted by chart review and by downloading ventilatory data from the ventilator. A registration of respiratory severity score will be done by a caregiver during the weaning period. This consists of a visual assessment of the work of breathing every 2 hours. For participants on NIV-NAVA consenting to the interventional part of the study a titration procedure will be conducted, afterwards serial electrical impedance tomography and lung and diaphragm ultrasound measurements will be done.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (< 37 weeks GA) supported with non-invasive respiratory support for at least 24 hours. Non-invasive respiratory support can consist of non-invasive NAVA, nasal continuous positive airway pressure (nCPAP) or high flow nasal canula (flow > 2 liters/min).The support can be given as primary respiratory support or as respiratory support after weaning from invasive ventilation (= after extubation).
* Infants can only be enrolled after written and signed informed consent by the parents.

Exclusion Criteria:

* Infant born after a gestational age of 37 weeks or more.
* Infants with major congenital malformations or chromosomal abnormalities (eg trisomy 18, congenital diaphragmatic hernia…)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Total duration of respiratory support | From birth until study completion, variating between 3 weeks and 3 months
  Total number of days of invasive and non-invasive respiratory support
Rate of bronchopulmonary dysplasia (BPD) or death | From birth until gestational age of 36 weeks
  Percentage of infants with BPD or death

SECONDARY OUTCOMES:
Duration of invasive respiratory support (days) | From birth until study completion, variating between 3 weeks and 3 months
Duration of non-invasive respiratory support (days) | From birth until study completion, between 3 weeks and 3 months
Description of mode of non-invasive respiratory support | From birth until study completion, between 3 weeks and 3 months
  Use of NIV-NAVA, CPAP, high flow nasal cannula, oxygen therapy
Use of surfactant and mode of administration | From birth until study completion, between 3 weeks and 3 months
Incidence of nosocomial infection | From birth until study completion, between 3 weeks and 3 months
Use of corticosteroids for the prevention or treatment of BPD | From birth until study completion, between 3 weeks and 3 months
  Use of any corticosteroid (systemic or local)
Length of hospital stay | From birth until study completion, between 3 weeks and 3 months
  Days of stay in the neonatal unit
Respiratory severity score (RSS) | From start of the weaning phase until respiratory support is stopped, up to 10 weeks
  RSS will be measured during the weaning phase of non-invasive respiratory support
NIV-NAVA breakpoint | At inclusion (within 24 hours)
  Definition of the breakpoint for patients of NIV-NAVA after following a prespecified titration protocol
Lung ultrasound score | At inclusion, day 3, day 7 and weekly thereafter as long as supported with NIV-NAVA, up to 10 weeks
  Lung ultrasound score will be scored at several time points
Diaphragm ultrasound | At inclusion, day 3, day 7 and weekly thereafter as long as supported with NIV-NAVA, up to 10 weeks
  Measurement of diaphragm thickness with ultrasound
Silent Spaces | At inclusion, day 3, day 7 and weekly thereafter as long as supported with NIV-NAVA as long as supported with NIV-NAVA, up to 10 weeks
  Parts (in % of global lung volume) of the lung that are not ventilated as measured with electrical impedance tomography (EIT)
Tidal volume (TV) | At inclusion, day 3, day 7 and weekly thereafter as long as supported with NIV-NAVA as long as supported with NIV-NAVA, up to 10 weeks
  Percentage of TV per 'Region of Interest' (ROI) as measured with electrical impedance tomography (EIT)
Center of Ventilation (CoV) | At inclusion, day 3, day 7 and weekly thereafter as long as supported with NIV-NAVA as long as supported with NIV-NAVA, up to 10 weeks
  As measured with electrical impedance tomography (EIT)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lefevere, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Filip Cools, PhD, Study Director — Universitair Ziekenhuis Brussel; Brenda Van Delft, Nurse, Study Chair — Universitair Ziekenhuis Brussel; Caitlin Jansen, Student, Study Chair — Vrije Universiteit Brussel; Lissa De Potter, MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Database on non-invasive ventilation has the potential to be shared but no concrete plan for sharing individual patient data is made.

REFERENCES:
- [Background] Baraldi E, Filippone M. Chronic lung disease after premature birth. N Engl J Med. 2007 Nov 8;357(19):1946-55. doi: 10.1056/NEJMra067279. No abstract available. PMID 17989387
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Lefevere J, Van Delft B, Vervoort M, Cools W, Cools F. Non-invasive neurally adjusted ventilatory assist in preterm infants with RDS: effect of changing NAVA levels. Eur J Pediatr. 2022 Feb;181(2):701-707. doi: 10.1007/s00431-021-04244-3. Epub 2021 Sep 17. PMID 34533644
- [Background] Harada E, Kinoshita M, Iwata S, Saikusa M, Tsuda K, Shindou R, Sahashi T, Kato S, Yamada Y, Saitoh S, Iwata O. Visual function scale for identification of infants with low respiratory compliance. Pediatr Neonatol. 2019 Dec;60(6):611-616. doi: 10.1016/j.pedneo.2019.02.006. Epub 2019 Mar 2. PMID 30905442
- [Background] Thomson J, Ruegger CM, Perkins EJ, Pereira-Fantini PM, Farrell O, Owen LS, Tingay DG. Regional ventilation characteristics during non-invasive respiratory support in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2021 Jul;106(4):370-375. doi: 10.1136/archdischild-2020-320449. Epub 2020 Nov 27. PMID 33246967
- [Background] Raimondi F, Yousef N, Migliaro F, Capasso L, De Luca D. Point-of-care lung ultrasound in neonatology: classification into descriptive and functional applications. Pediatr Res. 2021 Sep;90(3):524-531. doi: 10.1038/s41390-018-0114-9. Epub 2018 Jul 20. PMID 30127522
- [Background] Alonso-Ojembarrena A, Ruiz-Gonzalez E, Estepa-Pedregosa L, Armenteros-Lopez AI, Segado-Arenas A, Lubian-Lopez SP. Reproducibility and reference values of diaphragmatic shortening fraction for term and premature infants. Pediatr Pulmonol. 2020 Aug;55(8):1963-1968. doi: 10.1002/ppul.24866. Epub 2020 Jun 5. PMID 32458563